CLINICAL TRIAL: NCT05902507
Title: Magnetic Resonance Imaging in RadiotheRapy fOr bReast Cancer (MIRROR): A Pilot Study of MRI Simulation
Brief Title: Magnetic Resonance Imaging in Radiotherapy for Breast Cancer
Acronym: MIRROR
Status: Suspended | Type: Observational
Why Stopped: Operational delay, study to resume at later date
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: 22725; NCI-2023-03214 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast Cancer Participants: Participants will receive both MRI and CT simulation scans.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging Simulation

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging Simulation — Radiographic Image Simulation
  Other Names: MRI

SUMMARY:
This is a single-center, prospective pilot study evaluating feasibility and efficacy of incorporating magnetic resonance imaging (MRI) simulation into the planning of radiation treatment (RT) for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine feasibility of acquiring MRI simulation prior to RT planning.

EXPLORATORY OBJECTIVE:

I. To determine change in target volume with MRI simulation compared to Computerized tomography (CT) simulation.

OUTLINE: MRI simulation will be performed once at baseline. There is no follow up planned for study purposes. Patients will be followed as part of their regular clinical care.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with an Eastern Cooperative Oncology Group (ECOG) performance status <=2 (or Karnofsky ≥>=60%, see Appendix A).
2. Participants with the ability to understand and the willingness to sign a written informed consent document.
3. Participants may separately enroll on therapeutic clinical trials when they enroll on this trial. Note: All interventions on this protocol are standard of care, so enrollment on other therapeutic protocols is allowed at the discretion of the treating physician.
4. Patients must have pathologically confirmed invasive or in situ breast cancer.
5. Patients must have tumors in which adjuvant breast radiotherapy following breast conserving surgery is indicated, as determined by the treating physician.
6. Patients must be female. Note: Male patients are excluded due to the rarity of male breast cancer and difficulty in pursuing breast conserving surgery for male patients.

Exclusion Criteria:

1. Participants with a contraindication to MRI per the MRI checklist.
2. Patients with breast tumor or tumor bed not visualized at CT or MRI during RT planning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female participants with breast cancer planning to undergo breast conserving surgery (BCS) and RT outside of this protocol.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who completed scan | Day of MR imaging (1 day)
  Feasibility feasibility of acquiring MRI simulation prior to RT planning is defined as successfully acquiring MRI data at the specified time point in a participant's radiotherapy (RT) care plan

OTHER OUTCOMES:
Median absolute change in size of target | Day of MR imaging (1 day)
  To evaluate the absolute change in size of target based on CT data, versus with MRI data, the change in volume (measured in cubic centimeters (cc)) of the target with MRI simulation will be calculated compared to CT.
Median relative difference in size of target | Day of MR imaging (1 day)
  To evaluate the relative difference in size of target based on CT data, versus with MRI data, the change in volume (measured in cubic centimeters (cc)) of the target with MRI simulation will be calculated compared to CT.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Singer, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No